CLINICAL TRIAL: NCT00349362
Title: A Randomised Double Blind Placebo Controlled, Parallel Pilot Study to Test the Effect of Testosterone Replacement on Glycaemic Control and Arterial Wall Properties of Hypogonadal Men With Type 2 Diabetes Treated With Insulin
Brief Title: Testosterone for Men With Insulin Treated Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barnsley Hospital (Other)
Responsible Party: Prof Hugh Jones, Barnsley Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BDGH 264
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Hypogonadism; Diabetes
MeSH Terms: conditions — Hypogonadism; Diabetes Mellitus | interventions — Testosterone; Saline Solution

ARMS (2):
- Testosterone (Experimental): Testosterone injections- 200mg- every 2 weeks
  Interventions: Drug: Testosterone
- Placebo (Placebo Comparator): Normal saline injections- every two weeks
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Testosterone — Sustanon- 200mg intramuscular testosterone
  Arms: Testosterone
Drug: 0.9% saline — Saline intramuscular injection every two weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the effect of testosterone treatment on glycaemic control, arterial stiffness and IMT in hypogonadal men with type 2 diabetes treated with insulin.

DETAILED DESCRIPTION:
There is epidemiological data linking low serum testosterone levels in men with the development of diabetes. Clinical trials have indicated a potential benefit of testosterone treatment in improving diabetic control and insulin resistance. Type 2 diabetes is also associated with changes in arterial stiffness and IMT which are known to be linked to the presence of cardiovascular disease. Artificially induced hypogonadism results in increasing arterial stiffness whilst testosterone is known to improve risk factors for vascular disease and act as a vasodilator. The purpose of this pilot study is to test the effect of six months of testosterone replacement, given as testosterone esters 200mg from Sustanon 250 IM injection, on diabetes control in hypogonadal men with type 2 diabetes treated with insulin.

ELIGIBILITY:
Inclusion Criteria:

* males over 40 years old
* type 2 diabetes treated with insulin
* serum testosterone less than 12nmol/L on 2 consecutive morning samples
* symptoms attributable to hypogonadism

Exclusion Criteria:

* current or previous breast cancer
* current or previous prostate cancer
* raised prostate specific antigen or abdominal digital rectal examination suspicious of prostate cancer unless diagnosis excluded after specialist urology opinion and/or prostate biopsy
* severe symptoms of benign prostatic hypertrophy
* treatment with testosterone in the three months prior to the trial
* investigational drug treatment in the three months prior to the trial

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The effect of 6 months of testosterone replacement on diabetes control measured by HbA1c in hypogonadal men with type 2 diabetes treated with insulin. | 6 months

SECONDARY OUTCOMES:
The effect of testosterone on ultrasound measured intima-media thickness of the common carotid artery in the study population | 6 months
The effect of testosterone on male hypogonadism as assessed by the Ageing Males Symptoms (AMS) | 6 months
The effect of testosterone on markers of vascular risk; blood pressure, serum lipid levels, weight, waist circumference, body fat percentage, | 6 months
urinary micro-albumin, tumour necrosis factor alpha, and highly sensitive C reactive protein levels in the study population. | 6 months
The effect of the CAG repeat polymorphism in exon 1 of the androgen receptor gene on the response of the study population to testosterone. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Jones, BSc MD FRCP, Principal Investigator — Barnsley Hospital NHS Foundation Trust
Locations (1):
- Barnsley Hospital NHS Foundation Trust, Barnsley, South Yorkshire, United Kingdom